CLINICAL TRIAL: NCT03581773
Title: FASTERCC: Folic Acid Supplement Versus Placebo for Treating Mucositis Adverse Events in Metastatic Renal Cell Carcinoma Patients Receiving Targeted Therapy. A Randomized, Double-blind Trial From the Danish Renal Cancer Group (DARENCA Study-4)
Brief Title: Folic Acid Supplement Versus Placebo for Treating Mucositis Adverse Events in Metastatic Renal Cell Carcinoma Patients Receiving Targeted Therapy
Acronym: DARENCA4
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Niels Fristrup (Other)
Responsible Party: Sponsor-Investigator, Niels Fristrup, Principal Investigator, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FASTERCC
Record Dates: First submitted 2018-05-07; First posted 2018-07-10 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Mucositis; Stomatitis
MeSH Terms: conditions — Mucositis; Stomatitis | interventions — Folic Acid

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled phase II trial of the effectiveness of folic acid supplement for 12 weeks on mucositis. Both arms will receive best supportive care. No crossover is allowed.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The master randomization list will be created, maintained and kept in a locked, secure location at Hospitalsapoteket Region Midtjylland, Afdeling Herning. The randomization list will not be available to any person directly involved in the study, including the study centre personnel or the project team.
  Randomization will be performed via a central randomization service available in business hours on working days by fax 7843 5165. A block design randomization procedure will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment arm (Active Comparator): 5 mg of folic acid (1 tablet) per day for 12 weeks.
  Interventions: Drug: Folic Acid
- Placebo arm (Placebo Comparator): PLACEBO (1 tablet) per day for 12 weeks.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Folic Acid — 5 mg pr day for 12 weeks
  Arms: Treatment arm
Drug: Placebo Oral Tablet — 1 placebo pill pr day for 12 weeks
  Arms: Placebo arm

SUMMARY:
FASTERCC: Folic acid supplement versus placebo for treating mucositis adverse events in metastatic renal cell carcinoma patients receiving targeted therapy. A randomized, double-blind trial from the Danish renal cancer group (DARENCA study-4)

DETAILED DESCRIPTION:
Mucositis (nasal, oral, pharyngeal, anal, or genital) is often experienced in relation to TKI, immunotherapy or mTOR inhibitor treatment in mRCC patients.

The present trial will assess whether 12 weeks complementary treatment with folic acid in mRCC-patients receiving TKI- or mTOR inhibitor treatment or immunotherapy and displaying CTCAE mucositis grade ≥2 can reduce the degree of mucositis, compared to PLACEBO.

This is a randomized, double-blind, placebo-controlled phase II trial of the effectiveness of folic acid supplement for 12 weeks on mucositis. Both arms will receive best supportive care. No crossover is allowed.

The investigators anticipate a 96-month accrual period. The power calculation indicates a total of 50 patients per group are required.

Block randomization based on received TKI/ mTOR inhibitor/IT-treatment will be performed.

ELIGIBILITY:
Target population: Patients with inoperable, locally advanced, or metastatic renal cell carcinoma.

Inclusion Criteria:

1. Patients displaying CTCAE ≥2 mucositis during TKI, mTOR inhibitor or immunotherapy treatment.
2. Signed written informed consent obtained prior to any study specific procedures.
3. Patient must be willing and able to comply with the protocol.
4. Age ≥ 18.
5. Biopsy proven locally advanced or metastatic renal cell carcinoma.
6. Females with a negative serum pregnancy test unless childbearing potential can be otherwise excluded (postmenopausal, hysterectomy or oophorectomy) and not lactating.
7. Fertile women of childbearing potential (<2 years after last menstruation) and men must use effective means of contraception (oral contraceptives, intrauterine contraceptive device, barrier method of contraception in conjunction with spermicidal jelly or surgical sterilization).
8. Karnofsky Performance status ≥ 60%.

Exclusion Criteria:

1. Known hypersensitivity to folic acid.
2. Use of prednisolone more than 10 mg daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-12-20 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2028-12-20 (Estimated)

PRIMARY OUTCOMES:
CTCAE Mucositis | 16 weeks
  The degree of CTCAE mucositis (nasal, oral, pharyngeal, anal, or genital) according to the Common Terminology Criteria for Adverse Events v. 4.0 (CTCAE).

SECONDARY OUTCOMES:
PRO Mucositis frequency | 16 weeks
  The frequency of mucositis (nasal, oral, pharyngeal, anal, or genital) according to patient reported outcomes (PRO) by self assessment questionnaire using National Comprehensive Cancer Network Functional Assessment of Cancer Therapy Kidney Symptom Index-19 (NCCN-FACT FKSI-19) and a modified version of the M.D. Anderson Symptom Inventory (MDASI) for RCC.
Time to effect on mucositis | 16 weeks
  The median time to effect of study drug according to CTCAE 4.0 and PRO.
Dose reductions | 16 weeks
  The frequency of TKI/mTOR dose reductions in the two groups
Treatment discontinuations | 16 weeks
  The frequency of TKI/mTOR/immunotherapy treatment discontinuations in the two groups
Treatment withdrawals | 16 weeks
  The frequency of TKI/mTOR/immunotherapy treatment withdrawals in the two groups
GI adverse events degree | 16 weeks
  The degree of GI adverse events in the two groups according to CTCAE v. 4.0 and PRO.
Hand-foot syndrome degree | 16 weeks
  The degree of hand-foot syndrome in the two groups according to CTCAE v. 4.0 and PRO.
QOL NCCN | 16 weeks
  The quality of life in the two groups according to NCCN-FACT FKSI-19.
PRO Mucositis degree | 16 weeks
  The degree of mucositis (nasal, oral, pharyngeal, anal, or genital) according to patient reported outcomes (PRO) by self assessment questionnaire using National Comprehensive Cancer Network Functional Assessment of Cancer Therapy Kidney Symptom Index-19 (NCCN-FACT FKSI-19) and a modified version of the M.D. Anderson Symptom Inventory (MDASI) for RCC.
GI adverse events frequency | 16 weeks
  The frequency of GI adverse events in the two groups according to CTCAE v. 4.0 and PRO.
Hand-foot syndrome frequency | 16 weeks
  The frequency of hand-foot syndrome in the two groups according to CTCAE v. 4.0 and PRO.
QOL MDASI | 16 weeks
  The quality of life in the two groups according the M.D. Anderson Symptom Inventory for RCC.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Department of oncology, Aarhus, Central Region of Denmark
  - Department of Oncology, Herlev Hospital, Herlev

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Derived] Fristrup N, Donskov F. Folic Acid Reduces Mucositis in Metastatic Renal Cell Carcinoma Patients: A Retrospective Study. Clin Genitourin Cancer. 2019 Aug;17(4):254-259. doi: 10.1016/j.clgc.2019.03.023. Epub 2019 Apr 6. PMID 31101577